CLINICAL TRIAL: NCT00348387
Title: Immunogenicity and Safety of Imovax Polio in Chinese Infants Compared to Local OPV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IPV13
Record Dates: First submitted 2006-07-03; First posted 2006-07-04 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Poliomyelitis; Polio
Keywords: Imovax polio; poliomyelitis
MeSH Terms: conditions — Poliomyelitis | interventions — Poliovirus Vaccine, Inactivated; Poliovirus Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental)
  Interventions: Biological: Poliomyelitis Vaccine inactivated
- Group 2 (Active Comparator)
  Interventions: Biological: Poliomyelitis Vaccine in Dragee Candy (Human Diploid Cell)

INTERVENTIONS:
Biological: Poliomyelitis Vaccine inactivated — 0.5 mL, Intramuscular
  Other Names: IMOVAX Polio ™
  Arms: Group 1
Biological: Poliomyelitis Vaccine in Dragee Candy (Human Diploid Cell) — 1g dragee, oral
  Other Names: Poliomyelitis Vaccine in Dragee Candy
  Arms: Group 2

SUMMARY:
This study is intended to support the registration of IMOVAX Polio in China.

The primary objective of this Pase III trial is to compare IMOVAX Polio to the current Chinese standard of care (OPV) that is administered following a schedule of 2-3-4 months. The objective is to demonstrate that after the 3 doses primary series, in terms of seroprotection rates, IMOVAX Polio is not inferior to OPV. The safety of IPV will be assessed after each IPV dose.

ELIGIBILITY:
Inclusion Criteria:

* Aged 2 months (60-70 days) on the day of inclusion into the study
* Born at full term pregnancy ( over 36 weeks) with a birth weight ≥ 2.5 kg 2Ibs) or more
* Parent(s) or legal representative able to understand and give authorization and sign informed consent for participation
* Able to attend all planned clinic appointment and obey and follow all study instructions

Exclusion Criteria:

* Taking part in another clinical trial during the 4 weeks before the first trial vaccination
* Have plans to take part in another clinical trial d during this trial period
* Inborn or acquired decreased body natural defense, undertaking treatment that can reduce body's natural defense such as cancer drugs, radiation in the past six months or long term corticosteroid treatment
* Systemic reaction to any vaccine component or history of life-threatening reaction to study vaccine or any vaccine with the same ingredient(s)
* Prolonged or long time illness that could interfere with study or full participation
* Received blood or blood-derived products since birth
* Received any vaccine in the 4 weeks before the first trial vaccination is given (except BCG and hepatitis B)
* Have plans to receive any vaccine in the 4 weeks after the (or any) study vaccination is given (except DTacP)
* Previous vaccination against the poliomyelitis infection with the trial vaccine or another vaccine
* History of poliomyelitis infection (confirmed either by symptoms, blood or other laboratory test)
* Clinical or serological evidence of systemic illness including hepatitis B, hepatitis C or Human immunodeficiency virus (HIV)
* Bleeding disorder or a low platelet which do not allow vaccination into the muscle
* Had seizures in the past
* Febrile illness (axillary temperature ≥ 37.1°C) or acute illness on the day of inclusion

Ages: 60 Days to 70 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Actual)
Dates: Start 2006-06; Primary Completion 2008-09 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
To provide information concerning the immunogenicity of IMOVAX Polio™ vaccine | 1 month post-vaccination 3

SECONDARY OUTCOMES:
To provide information concerning the safety of IMOVAX Polio™ vaccine | Entire study period

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (2):
- China (2):
  - Guilin
  - PingLe County

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com